CLINICAL TRIAL: NCT03330392
Title: An 8 Week, Randomized, Double-blind, Placebo-controlled Clinical Trial of AGP on Immune Enhancing Effects
Brief Title: Evaluation of Efficacy and Safety of AGP on Immune Enhancement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Principal Investigator, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CTCF2_2017_AGP
Record Dates: First submitted 2017-10-31; First posted 2017-11-06 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Immune Function

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AGP (Experimental): take two tablets per day (500 mg/day) for 8 weeks.
  Interventions: Dietary Supplement: AGP
- Placebo (Placebo Comparator): take two tablets per day for 8 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: AGP — take two tablets per day (500 mg/day) for 8 weeks
  Arms: AGP
Dietary Supplement: Placebo — take two tablets per day (500 mg/day) for 8 weeks
  Arms: Placebo

SUMMARY:
The researchers investigated the immune enhancing effects of AGP for Korean participants.

DETAILED DESCRIPTION:
The aim of the study is to investigate the effects of AGP on immune enhancement based on 8 week, randomized, double-blind, placebo-controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* The levels of white blood cells within range 3x10^3/μL~8x10^3/μL
* have had at least two cold in the last 12 months.

Exclusion Criteria:

* subjects with BMI<18.5 kg/m^2
* subjects taking medications such as immune related drug or functional foods
* history of disease that could interfere with the test products or impede their absorption
* pregnant or lactating women and heavy smokers.
* being judged by the responsible physician of the local study center as unfit to participate in the study

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-09-07 (Actual); Study Completion 2017-10-27 (Actual)

PRIMARY OUTCOMES:
Natural killer cell activity | 0 week, 8 week
  Changes of NK cell activity were assessed before and after the intervention.

SECONDARY OUTCOMES:
Interleukin-1β | 0 week, 8 week
  Changes of IL-1β were assessed before and after the intervention.
Interleukin-6 | 0 week, 8 week
  Changes of IL-6 were assessed before and after the intervention.
Interleukin-12 (IL-12) | 0 week, 8 week
  Changes of IL-12 were assessed before and after the intervention.
Interferon-γ (IFN-γ) | 0 week, 8 week
  Changes of IFN-γ were assessed before and after the intervention.
Tumor necrosis factor-α (TNF-α) | 0 week, 8 week
  Changes of TNF-α were assessed before and after the intervention.
Changes of White blood cell (WBC) | 0 week, 8 week
  Changes of WBC were assessed before and after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center for Functional Foods Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea